CLINICAL TRIAL: NCT06168513
Title: Developing a Real-Time PCR Assay for Fusobacterium and Epidemiological Analysis of Tumor Patients
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Hongwei Zhou, Professor, Zhujiang Hospital
Other Study IDs: ZhujiangHstt
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Fusobacterium Infections
Keywords: Fusobacterium; PCR
MeSH Terms: conditions — Fusobacterium Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: The inclusion criteria for this study encompassed fecal specimens obtained from patients with a documented history of tumor, specifically those who received their primary or initial tumor diagnosis at our hospital.
- Healthy control: (1) Individuals who were in good health, devoid of evident diseases, and possessed normal physical examination reports; (2) Individuals who had not experienced significant chronic illnesses, such as hypertension, diabetes, chronic kidney disease, etc., in recent years, in order to exclude those who had been unwell but had normal physical examination reports; (3) Age and gender were matched with the case group.

SUMMARY:
This study presents an academic approach to developing a fluorescence quantitative PCR detection method capable of accurately measuring the presence of Fusobacterium (specifically F. nucleatum, F. mortiferium, F. varium, F. ulcerans, F. and F. necrogens) in human fecal samples. It aims to perform an epidemiological analysis on the presence of Fusobacterium in patients with tumors, elucidating the prevalence of Fusobacterium members in this patient population. Additionally, it seeks to investigate the potential correlation between Fusobacterium presence and various test indicators, diagnostic predictions, and prognosis outcomes.

DETAILED DESCRIPTION:
Fusobacterium nucleatum, a gram-negative obligate anaerobic bacterium, is known to colonize the oral cavity and is implicated in various diseases affecting the oropharynx, gastrointestinal tract, cardiovascular vessels, and genital tract. Precise classification of the Fusobacterium genus is of utmost importance as it will facilitate a deeper understanding of the pathogenicity of its members in tumor development, establish an accurate etiological association with tumors, and ultimately enhance clinical practice and epidemiological investigations.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for this study encompassed fecal specimens obtained from patients with a documented history of tumor, specifically those who received their primary or initial tumor diagnosis at our hospital.
* Inclusion criteria for the control group consisted of the following: (1) Individuals who were in good health, devoid of evident diseases, and possessed normal physical examination reports; (2) Individuals who had not experienced significant chronic illnesses, such as hypertension, diabetes, chronic kidney disease, etc., in recent years, in order to exclude those who had been unwell but had normal physical examination reports; (3) Age and gender were matched with the case group.

Exclusion Criteria:

The exclusion criteria for this study include: A) Individuals who have taken an antimicrobial preparation within the past three months. B) Samples that lack complete information and cannot be traced back to their source. C) Samples with an insufficient volume for detection. D) Samples that do not meet the requirements for sample collection and preservation.

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The inclusion criteria for this study encompassed fecal specimens obtained from patients with a documented history of tumor, specifically those who received their primary or initial tumor diagnosis at our hospital.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Fusobacterium | baseline
  Fusobacterium in stool detected using PCR

CONTACTS AND LOCATIONS:
Overall Officials: Houwei Zhou, professor, Study Chair — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No